CLINICAL TRIAL: NCT04817475
Title: Live Stream of Prehospital point-of Care Ultrasound During Cardiopulmonary Resuscitation
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Hafner, Clinical Investigator, Medical University of Vienna
Other Study IDs: 2410/2020
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cardiopulmonary Resuscitation; Echocardiography; Ultrasound
Keywords: Ultrasound diagnstics; Prehospital emergency medicine; Telemedicine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Point-of-care ultrasound with tele-supervision: Point-of-care ultrasound of patients with a out-of-hospital cardiac arrest will be performed with tele-supervision.
  Interventions: Other: Point-of-care ultrasound with tele-supervision

INTERVENTIONS:
Other: Point-of-care ultrasound with tele-supervision — Point-of-care ultrasound of patients with a out-of-hospital cardiac arrest will be performed with tele-supervision.

SUMMARY:
Background: Point-of-care ultrasound (POCUS) has been suggested as a useful tool in out-of-hospital cardiac arrest (OHCA) for diagnosis and treatment of reversible causes. However, in prehospital emergency medicine performing ultrasound and the translation of the findings can be challenging. As new prehospital ultrasound devices offer the possibility for remote supervision, the impact of tele-supervision on the performance of POCUS during OHCA is unclear.

Aims: This prospective observational study aims to evaluate if POCUS with tele-supervision can be performed during CPR without any additional hands-off periods longer than 5 seconds.

Methods: In total 30 patients with OHCA, where POCUS is considered, will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

Patients with prehospital cardiac arrest, where POCUS is considered during cardiac pulmonary resuscitation, will be included.

Exclusion Criteria:

* under the age of 18,
* if POCUS is not considered or if POCUS will lead to a delay of live-saving treatment or transportation.
* pregnant patients
* patients with a body-mass-index (BMI) above 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 critically ill patients suffering from acute cardiopulmonary resuscitation will be included in this study. POCUS will be performed with tele-supervision.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Hands-off time during prehospital cardiopulmonary resuscitation | through study completion, an average of 1 year
  The primary outcome of this study evaluates, if POCUS with tele-supervision can be performed during prehospital cardiopulmonary resuscitation without any additional hands-off period longer than 5 seconds

SECONDARY OUTCOMES:
Impact of real-time supervision of POCUS during cardiopulmonary resuscitation on the duration time of POCUS | through study completion, an average of 1 year
  Impact of real-time supervision of POCUS during cardiopulmonary resuscitation on the duration time of POCUS
Impact of real-time supervision of POCUS during cardiopulmonary resuscitation on changing of diagnosis of suspected cause of out-of-hospital cardiac arrest. | through study completion, an average of 1 year
  Impact of real-time supervision of POCUS during cardiopulmonary resuscitation on changing of diagnosis of suspected cause of out-of-hospital cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: Department of Anaesthesia & General Intensive Care, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Anaesthesia & General Intensive Care, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hafner C, Manschein V, Klaus DA, Schaubmayr W, Tiboldi A, Scharner V, Gleiss A, Thal B, Krammel M, Hamp T, Willschke H, Hermann M. Live stream of prehospital point-of-care ultrasound during cardiopulmonary resuscitation - A feasibility trial. Resuscitation. 2024 Jan;194:110089. doi: 10.1016/j.resuscitation.2023.110089. Epub 2023 Dec 16. PMID 38110144